CLINICAL TRIAL: NCT07045402
Title: The Effect of Kangaroo Care and Maternal Voice on Comfort, Anthropometric Measurements, and Transition to Oral Feeding in Preterm Infants
Brief Title: Effect of Developmental Care on Comfort, Growth, and Oral Feeding Transition in Preterm Infants
Acronym: KCareInfant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Negarin Akbari, Assisstant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4507
Record Dates: First submitted 2025-06-04; First posted 2025-07-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Infant, Premature; Kangaroo Mother Care; Comfort; Feeding; Oral Feeding Performance; Facilitated Tucking
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kangaroo Care + Maternal Voice + Fetal Position Group (Experimental): Infants in this group, once clinically stable, will receive kangaroo care with their mothers for one hour, at least five days a week, immediately after their enteral feeding until they transition to full oral feeding. During the first 15 minutes of skin-to-skin contact, the mother will tell a story to the infant. After the kangaroo care, the infants will be placed in an incubator, and a lateral fetal position will be maintained for half an hour. During this process, no intervention will be made unless necessary.
  Until the infant transitions to full oral feeding, comfort will be assessed once a day, at least five days a week, using the Neonatal Comfort Behavior Scale: before feeding, immediately before finishing kangaroo care (at 60 minutes), and 30 minutes after the fetal position (at 90 minutes). On the days kangaroo care is applied, before feeding, the infant will be weighed using a ±10-gram sensitive digital baby scale, and their length and head circumference will be measured with
  Interventions: Other: Kangaroo Care + Maternal Voice + Fetal Position Group
- Control Group: (Fetal Position group) (Active Comparator): Infants in this group, whose mothers are unavailable, will receive only lateral fetal positioning for one and a half hours immediately after their enteral feeding, at least five days a week, until they transition to full oral feeding, in the incubator.
  Until the infant transitions to full oral feeding, the same measurements will be taken and recorded as those for the Kangaroo Group.
  Interventions: Other: control group

INTERVENTIONS:
Other: Kangaroo Care + Maternal Voice + Fetal Position Group — After ethical approval, all infants with a gestational age between 30-34 weeks in Neonatal Intensive Care Unit will be assessed. Parents of eligible infants will be informed about the study and asked to provide written consent. The infants will then be assigned to one of two groups: kangaroo care + mother's voice + fetal position (n=34) or fetal position only (n=34). In the first group, after tube feeding, infants will receive one hour of kangaroo care with the mother, including reading a story for the first 15 minutes. After finishing kangaroo care,they will then be placed in a fetal position in an incubator for 30 minutes. Comfort levels, weight, length, and head circumference will be measured daily until oral feeding begins, and the impact of kangaroo care and the mother's voice on the transition to full oral feeding will be assessed. All procedures will occur between 08:00 and 16:00.
  Arms: Kangaroo Care + Maternal Voice + Fetal Position Group
Other: control group — After ethical approval, all infants with a gestational age between 30-34 weeks in the Neonatal Intensıve Care Unit will be assessed. Parents of eligible infants will be informed about the study and asked to provide written consent. If infant is in the fetal position group, after being fed by a oral gastric tube, they will be placed in an incubator and positioned in a fetal position similar to that in the womb for one and a half hours. During all these procedures, infant's comfort levels will be assessed using a scale (form), and their weight, length, and head circumference will be measured every morning until they begin oral feeding. Additionally, the effect of the fetal position on infant's transition to full oral feeding will be evaluated.All procedures will take place between 08:00 and 16:00.
  Arms: Control Group: (Fetal Position group)

SUMMARY:
This randomized controlled study aims to evaluate the effects of kangaroo care combined with maternal voice and fetal positioning on the comfort, growth, and transition to full oral feeding in preterm infants aged 30 to 34 weeks gestation. After ethical approval, eligible infants in the neonatal clinic will be randomly assigned to either the intervention group receiving kangaroo care, maternal voice, and fetal positioning, or a control group receiving only fetal positioning in the incubator. The intervention involves daily one-hour kangaroo care sessions with maternal storytelling, followed by positioning in the lateral fetal posture, continuing at least five days per week until infants achieve full oral feeding. Infant comfort will be assessed regularly using the Neonatal Comfort Behavior Scale before feeding, immediately after kangaroo care, and after fetal positioning. Growth parameters, including weight, length, and head circumference, will be measured and recorded on kangaroo care days. The control group will receive routine fetal positioning without kangaroo care, with identical measurements taken. The study aims to determine whether kangaroo care combined with maternal voice and fetal positioning improves infant comfort, supports growth, and facilitates the transition to full oral feeding in preterm newborns.

DETAILED DESCRIPTION:
After obtaining ethical approval for the study, all infants with a gestational age between 30 and 34 weeks in the Neonatal Clinic will be evaluated. After the infants are assigned to groups, the data collection phase will begin.

Before data collection, the researcher will provide necessary information about the study to the families of eligible newborns and answer their questions. Infants whose parents give written consent to participate will be included in the study. Information on the newborn and parent introductory information form will be recorded by the researcher. All procedures will be conducted between 08:00 and 16:00.

**Group 1: Infants Receiving Kangaroo Care (Kangaroo Care + Mother's Voice + Fetal Position Group):** Infants in this group, once clinically stable, will receive kangaroo care with their mothers for one hour immediately after enteral feeding at least five days a week until they transition to full oral feeding. During the first 15 minutes of skin-to-skin contact, the mother will read a story to the baby. After kangaroo care, infants will be placed in the incubator and positioned in the lateral fetal position for half an hour. During this process, interventions will be minimized unless necessary.

Until full oral feeding is achieved, comfort will be assessed using the Neonatal Comfort Behavior Scale at least five days a week, once daily: before feeding, immediately before ending kangaroo care (at 60 minutes), and 30 minutes after fetal positioning (at 90 minutes).

On the mornings of kangaroo care days, before feeding, the infant's growth will be evaluated: the infant will be weighed naked using a digital baby scale sensitive to ±10 grams; length and head circumference will be measured with a non-stretchable measuring tape and recorded.

**Group 2: Control Group (Fetal Position Group):** Infants in this group, whose mothers are not able to attend, will be placed in the incubator in the lateral fetal position for one and a half hours immediately after enteral feeding at least five days a week until full oral feeding is achieved.

The same measurements performed in the Kangaroo Care Group will be conducted and recorded for infants in this group until full oral feeding transition.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with a gestational age between 30-34 weeks.
2. The mother's ability to read and write.
3. The infant must be fully enterally fed at the time of enrollment in the study.
4. Infants who are being fed via orogastric tube at the time of enrollment.
5. Infants whose mothers agree to engage in skin-to-skin contact for 1 hour, five sessions per week, with auditory stimulation (storytelling) for 15 minutes will be included in the study.
6. Infants whose mothers cannot participate in the study (due to health issues or other reasons) or refuse kangaroo care will be placed in the control group, where routine service care will be applied.

Exclusion Criteria:

1. Presence of a congenital anomaly or genetic disease.
2. Requirement of ventilator support.
3. Infants receiving antibiotics for sepsis or suspected sepsis.
4. Administration of sedative treatment.
5. Having an intracranial hemorrhage greater than grade II.
6. The mother having a physical condition that prevents skin-to-skin contact.
7. The mother using substances or alcohol.

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Comfort | Until full oral feeding is achieved, evaluations will be conducted at least five days a week, once a day, at the following time points: before feeding, immediately before ending kangaroo care (at the 60th minute), and 30 minutes after placing the infant.
  The scale is a Likert-type tool developed to assess the sedation and comfort needs, as well as pain and distress levels, of newborns monitored in intensive care units. The Numeric Rating Scales are based on the caregiver nurse's observations. Each item on the scale is scored from 1 to 5, and the total score is used for evaluation. The minimum possible score on the Neonatal Comfort Behavior Scale is 6, and the maximum is 30. A total score between 9 and 13 indicates that the infant is comfortable, while a score between 14 and 30 suggests that the infant is experiencing pain or distress, is uncomfortable, and requires comfort-providing interventions.
Transition to Oral Feeding | From the date of study enrollment until the date of transition to full oral feeding, assessed for up to 8 weeks.
  The time from the infant's inclusion in the study until the transition to full oral feeding will be evaluated.

SECONDARY OUTCOMES:
Anthropometric measurements | From the first day of the intervention until the end of the 4-week study period, measurements will be taken at 9:00 a.m. prior to feeding on each day kangaroo care is provided.
  On the mornings of the days when kangaroo care will be applied, the infant's growth and development will be assessed before feeding. The baby will be weighed naked using a digital baby scale with ±10 grams sensitivity. Body length and head circumference will be measured using a non-flexible measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Canan GENÇ, Ph.D student, Principal Investigator — Fenerbahce University; Duygu Gözen, Ph.D, Study Chair — Koç University; NEGARIN Akbari, Ph.D, Study Chair — Fenerbahce University; Melek Selalmaz, Ms.c, Principal Investigator — ŞİŞLİ HAMİDİYE ETFAL TRAINING AND RESEARCH HOSPITAL; Ali Bulbul, Doctor, Principal Investigator — ŞİŞLİ HAMİDİYE ETFAL TRAINING AND RESEARCH HOSPITAL
Locations (1):
- Fenerbahce University, Istanbul, Turkey (Türkiye)